CLINICAL TRIAL: NCT07284277
Title: Phase Ib-II, Non-randomized, Open-label Study of Tumor Treating Fields (TTFields, 150 kHz) Concomitant With modFOLFIRINOX for Front-line Treatment of Metastatic Pancreatic Adenocarcinoma (NOVOFFOX)
Brief Title: TTFields and Chemotherapy in Metastatic Pancreatic Adenocarcinoma (mPDAC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOVOFFOX; 2024-511459-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Adenocarcinoma Metastatic; Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Cancer; Metastatic Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, open-label, one arm, multi-center study of the combination of NovoTTF-200T system with modFOLFIRINOX.
  A safety run in cohort of six patients will be conducted to assess toxicity and safety of the combination. Then, a second part consisting of an expansion cohort in which the rest of accorded patients will be performed.
  The study shall end when the final randomized patient has completed the study, all the planned visits have been carried out and any inconsistencies have been resolved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TTFields concomitant with modFOLFIRINOX (Experimental): Patients will receive a combination of modFOLFIRINOX with TTFields (150 kHz) in 14-day cycles.
  Interventions: Combination Product: TTFields concomitant with modFOLFIRINOX

INTERVENTIONS:
Combination Product: TTFields concomitant with modFOLFIRINOX — Patients will receive the following medication in 14-day cycles:
  ModFOLFIRINOX
  * Folic acid (Leucovorin) 400mg/m2 (D,L, racemic form) or 200mg/m2 (L-isomer form)
  * 5-fluorouracil (5Fu) 2400 mg/m2
  * Oxaliplatin 85mg/m2
  * Irinotecan 150-180mg/m2
  Combined with TTFields, which is a portable battery operated system intended for continuous home use (at least 18h/day) which delivers TTFields at a frequency of 150kHz to produces electric forces intended to disrupt cancer cell division.

SUMMARY:
The purpose of this clinical trial is to assess the safety and tolerability of TTFields in combination with chemotherapy in adults with metastatic pancreatic adenocarcinoma based on treatment-emergent adverse events of chemotherapy (modFOLFIRINOX) or device (TTFields).

The main questions it aims to answer are:

* Is TTFields treatment safe for the patients in combination with modFOLFIRINOX?
* Are participants compliant with the treatment?
* Is Is TTFields treatment effective in combination with modFOLFIRINOX against metastatic pancreatic adenocarcinoma?

DETAILED DESCRIPTION:
This is a phase Ib-II, non-randomized, open-label, one arm, multi-center study of the combination of NovoTTF-200T system with modFOLFIRINOX for the evaluation of the safety of the treatment in patients with metastatic pancreatic adenocarcinoma.

Pancreatic ductal adenocarcinoma (PDAC) is the eight cause of cancer mortality in men and ninth in women worldwide. Nearly 50,000 patients are diagnosed annually and almost all of them are expected to die from the disease without any challenges in survival in the last decade. Unfortunately, in most of the cases the disease is already disseminated when tumor related symptoms appear, with 5-year survival rate of less than 8 percent in this population (Siegel et al, 2020).

Tumor Treating Fields (TTFields) are a non-invasive regional antimitotic treatment with minimal toxicity. TTFields act by delivering alternate low-intensity electric fields (1-3 V/cm), intermediate frequency (100-300 kHz), and alternating electric fields to the tumor using non-invasive transducer arrays placed on the skin around the region of the body containing the tumor. TTFields act predominantly during two phases of mitosis: 1) during metaphase, by disrupting the formation of the mitotic spindle; and 2) during cytokinesis, by dielectrophoretic dislocation of intracellular constituents, leading apoptosis.

There is an increasing interest in the addition of immunotherapy to treatment pancreatic adenocarcinoma. Thus, combining TTFields with immunotherapy represents an interest for future clinical trials. However, the combination of TTFields with FOLFIRINOX chemotherapy scheme has not been evaluated yet. In this trial, it is proposed to evaluate the combination of TTFields with modFOLFIRINOX chemotherapy in metastatic PDAC patients with liver metastases. The aim is to analyze both the safety of combining TTFields with modFOLFIRINOX chemotherapy scheme, and to study the potential effect of TTFields and chemotherapy on the TME of liver metastasis.

Each patient shall participate in the trial for a maximum of 24 months. The trial will consist in two consecutive parts:

* A first part (Phase Ib) consisting of a safety run-in cohort: This first part will include 6 patients that will be treated with standard dose of modFOLFIRINOX scheme combined with TTFields.
* A second part (Phase II) consisting of an expansion cohort in which the rest of accorded patients will be included.

ELIGIBILITY:
Inclusion Criteria:

All the patients should comply with the following criteria for inclusion:

1. Histological/cytological diagnosis of pancreatic adenocarcinoma.
2. The patient should be 18 years of age and older.
3. The patient has given consent to participate in the study.
4. The patient should be able to comply with all the requirements of the clinical trial.
5. Life expectancy of at least 3 months.
6. Metastatic disease with, at least, one hepatic lesion that must be accessible for biopsy.
7. Measurable disease as defined by Response Evaluation Criteria in Solid Tumor v1.1 (RECIST 1.1) apart from the liver lesion to be biopsied.
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
9. Amenable and assigned by the investigator to receive therapy with modFOLFIRINOX.
10. Prior chemotherapy or radiotherapy on the neoadjuvant or adjuvant setting is allowed as long as at least six months have elapsed since last chemotherapy treatment.
11. Able to operate the Novo TTF-200T System independently or with the help of a caregiver.
12. Adequate hematologic and organ function, defined by the following laboratory test results, obtained during the screening period and before C1D1.

    1. WBC higher than or equal to 2.5 x 10^9/L.
    2. ANC higher than or equal to 1.5 x 10^9/L without granulocyte colony-stimulating factor support.
    3. Platelet count higher than or equal to 100 x 10^9/L without transfusion.
    4. Hemoglobin higher than or equal to 9 g/dL. Patients may be transfused to meet this criterion.
    5. Albumin higher than or equal to 2.5 g/dL.
    6. Serum bilirubin lower than or equal to 1.5 times the upper limit of normal (ULN); patients with known Gilbert´s disease may have a bilirubin value lower than or equal to 3 x ULN.
    7. INR and aPTT lower than or equal to 1.5 x ULN.
    8. AST, ALT, lower than or equal to 5 x ULN.
    9. Serum creatinine lower than or equal to 1.5 x ULN or Creatinine Clearance higher than or equal to 30ml/min (calculated using Cockcroft-Gault formula).
13. For women of childbearing potential: Negative serum pregnancy test within 14 days prior to C1D1. Agreement to remain abstinent (refrain from heterosexual intercourse) or use of contraceptive methods that result in a failure rate of lower than or equal to 1 percentage per year during the treatment period (combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal o transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable o implantable); intrauterine device (IUD) or intrauterine hormone-releasing system (IUS); bilateral tubal occlusion or vasectomized partner) and for at least 180 days after the last study treatment. A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (higher than or equal to 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).

Exclusion Criteria:

Patients who present any of the following criteria for exclusion cannot be included in the clinical trial:

1. Malignancies other than pancreatic cancer within 3 years prior to Cycle 1 Day 1 (C1D1) with the exceptions of those with a negligible risk of metastasis or death (e.g., expected 5-year overall survival higher than 90 percentage), treated with expected curative outcome (such as but not limited to: adequately treated in situ carcinoma of the cervix, basal squamous or melanomatous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ of the breast treated surgically with curative intent).
2. Previous treatment with chemotherapy for metastatic pancreatic ductal adenocarcinoma.
3. Untreated CNS metastases. Treatment of brain metastases, either by surgical or radiation techniques, must have been completed at least 4 weeks prior to study entry.
4. Known dihydropyrimidine dehydrogenase deficiency or thymidylate synthase gene polymorphism predisposing the patient for 5-fluorouracil (5-FU) toxicity.
5. Previous radiation therapy within 14 days prior to C1D1 and/or persistence of radiation-related adverse effects.
6. Implantable electronic medical devices in the torso, such as pacemakers.
7. Known severe hypersensitivities to medical adhesives or hydrogel, or history of severe allergic, anaphylactic, or other hypersensitivity reactions to any of the study treatments used.
8. Spinal cord compression not definitively treated with surgery and/or radiation.
9. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.
10. Pregnant and lactating women
11. Patients who have received brivudine, sorivudine or analogues 4 weeks prior to Fluoracile administration.
12. Serious co-morbidities, including but not limited to:

    1. History of significant cardiovascular disease unless the disease is well controlled. Significant cardiac disease includes second/third degree hart block; significant ischemic heart disease; poorly controlled hypertension; congestive heart failure of the New York Heart Association (NYHA) Class II or worse.
    2. History of cerebrovascular accident (CVA) within 3 months prior to randomization or that is not stable.
    3. Active infection or serious underlying medical condition that would impair the ability of the patient to receive protocol therapy.
    4. History of any psychiatric condition that might impair patient´s ability to understand or comply with the requirements of the study or to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile in patients with mPDAC treated at 1L with TTFields concomitantly with modFOLFIRINOX | From the beginning of the first treatment cycle (cycle 1; each treatment cycle is 14 days) through study completion (for a maximum of 24 months per patient since inclusion)
  Toxicity profile measured by the rate of patients with treatment-emergent adverse events (TEAEs), using CTCAE v5.0

SECONDARY OUTCOMES:
Total hours with TTField device functioning during every 14 days chemotherapy cycle | From the beginning of the first treatment cycle (cycle 1; each treatment cycle is 14 days) until discontinuation of last study treatment (for a maximum of 24 months per patient since inclusion).
  Total account of hours with TTField device functioning during every 14days chemotherapy cycle in the ITT population.
Quality of life (QoL) assessment | Screening visit, from cycle 13 (since completion of treatment with mFOLFIRINOX) onwards at each visit with test according to protocol, and at post-treatment termination visit (for a maximum of 24 months per patient since inclusion).
  Quality of life assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire of 30 items (EORTC QLQ-30). Questions 1-28: scale from 1 to 4, where 1 means a better quality of life and 4 indicates a worse quality of life; questions 29-30: scale from 1 to 7, where low scores indicate poorer health and quality of life, while high scores indicate better health and quality of life.
Progression-free survival (PFS) | Every 8 weeks from the beginning of the first treatment cycle (cycle 1) through study completion (for a maximum of 24 months per patient since inclusion).
  The time in months from first modFOLFIRINOX administration until disease progression based on CT scan collected on the study according to RECIST 1.1 criteria or any cause related death, whichever occurs first.
Overall survival (OS) | Since inclusion through study completion (for a maximum of 24 months per patient since inclusion).
  The time from first modFOLFIRINOX administration until patient death (if it occurs).
Overall response rate (ORR) | Every 8 weeks from the beginning of the first treatment cycle (cycle 1) through study completion (for a maximum of 24 months per patient since inclusion).
  The percentage of patients with complete response (CR) or partial response (PR) as best overall response (BOR) according to RECIST 1.1.
Disease control rate (DCR) | Every 8 weeks from the beginning of the first treatment cycle (cycle 1) through study completion (for a maximum of 24 months per patient since inclusion).
  The percentage of patients with CR or PR and the percentage of subjects with stable (SD) of at least 12 weeks duration as BOR according to RECIST 1.1.
Treatment impact on T-cell populations in the tumor and/or tumor periphery | At cycle 1 day 1 (each treatment cycle is 14 days), cycle 2 day 1, and cycle 5 day 1, and after discontinuation of last study treatment until disease progression (for a maximum of 24 months per patient since inclusion).
  Exploratory analyses on T-cell populations may include but will not be limited to Tumor-infiltrating lymphocytes (TILS) percentage measurement (immunohistochemistry (IHC)), percentage of different T-cell populations (e.g. CD8 or CD3) and RNAseq (antitumoral gene signatures evaluation), PD1-PDL1 expression (IHC).
Treatment impact on the immunosuppressive myeloid cells in the TME and peripheral blood: | At cycle 1 day 1 (each treatment cycle is 14 days), cycle 2 day 1, and cycle 5 day 1, and after discontinuation of last study treatment until disease progression (for a maximum of 24 months per patient since inclusion).
  Exploratory analyses on myeloid cells may include but will not be limited to RNAseq (immunosuppressive gene signature evaluation) and cytometry (changes on peripheral blood mononuclear cells).
Exploratory microbiome analysis | At screening, cycle 2 day 1 (each treatment cycle is 14 days), and cycle 5 day 1, and after discontinuation of last study treatment until disease progression (for a maximum of 24 months per patient since inclusion).
  Evaluation of microbiome communities via metagenomics sequencing in stool samples and identification of bacterial-derived metabolites in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Ponz Sarvisé, MD, PhD, Principal Investigator — Clínica Universidad de Navarra; Patricia Seoane Couselo, MD, Principal Investigator — Hospital Universitario de Araba; Fernando Garicano Goldáraz, MD, Principal Investigator — Hospital de Galdakao; Alberto Muñoz Llarena, MD, Principal Investigator — Hospital Universitario de Cruces; Ángela Lamarca Lete, MD, PhD, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (5):
- Spain (5):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Fundación Jiménez-Díaz, Madrid
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Álava

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949